CLINICAL TRIAL: NCT00038428
Title: Phase 2 Study of TLK286 in Platinum Resistant Advanced Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, M.D. Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2003
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-06

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — TER 286

INTERVENTIONS:
Drug: TLK286

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of TLK286 given intravenously once every week in the treatment of patients with advanced ovarian cancer that is resistant to platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Histologic diagnosis of ovarian cancer
* Recurrent or persistent disease following primary therapy
* Measurable disease
* Prior treatment with at least one but no more than three prior chemotherapy regimens
* Resistant or refractory to platinum-based chemotherapy
* At least 18 years of age
* Good performance status (ECOG 0 to 1)
* Adequate liver, renal and bone marrow function

Exclusion criteria

* Pregnant or currently breast feeding
* Treatment with chemotherapy or immunotherapy within four weeks
* Prior radiation to the whole pelvis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-06; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas